CLINICAL TRIAL: NCT01387490
Title: The Effect of Telephone Follow up on Outcome for Service Members With Mild TBI/PTSD
Brief Title: CONcussion Treatment After Combat Trauma (CONTACT)
Acronym: CONTACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTRuST-CONTACT
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury; Telephone counseling
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized Scheduled Telephone Support (ISTS) (Experimental): ISTS is a telephone intervention that provides injury-related education, training in problem solving, and focused behavioral strategies for problems (e.g., anxiety, depression) that commonly co-occur with Mild Traumatic Brain Injury (MTBI). ISTS also includes access to usual care and web-based and printed educational material. The 12 phone calls included in ISTS will be administered over a 6-month period.
  Interventions: Behavioral: Individualized Scheduled Telephone Support (ISTS)
- Usual Care (UC) (Other): UC is the usual care provided to service members attending the Traumatic Brain Injury (TBI) Clinics at Madigan Army Medical Center and Womack Army Medical Center, plus web-based education and 12 mailings of educational materials over a 6-month period.
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Behavioral: Individualized Scheduled Telephone Support (ISTS) — ISTS is a telephone intervention that provides injury-related education, training in problem solving, and focused behavioral strategies for problems (e.g., anxiety, depression) that commonly co-occur with Mild Traumatic Brain Injury (MTBI). ISTS also includes access to usual care and web-based and printed educational material. The 12 phone calls included in ISTS will be administered over a 6-month period.
  Arms: Individualized Scheduled Telephone Support (ISTS)
Other: Usual Care (UC) — UC is the usual care provided to service members attending the Traumatic Brain Injury (TBI) Clinics at Madigan Army Medical Center and Womack Army Medical Center, plus web-based education and 12 mailings of educational materials over a 6-month period.
  Arms: Usual Care (UC)

SUMMARY:
This study compares the effects of Individualized Scheduled Telephone Support (ISTS) and Usual Care (UC) for service members with Mild Traumatic Brain Injury (mTBI). A total of 400 service members will participate in this study. ISTS is a telephone intervention that provides injury-related education, training in problem solving, and focused behavioral strategies for problems (e.g. anxiety, depression) that commonly co-occur with MTBI. ISTS also includes access to usual care and web-based and printed educational material. The 12 phone calls included in ISTS will be administered over a 6-month period. UC is the usual care provided to service members attending the Traumatic Brain Injury (TBI) Clinics at Madigan Army Medical Center and Womack Army Medical Center, plus web-based education and 12 mailings of educational materials over a 6-month period. Subjects will complete major assessments at study entry and then 6 months and 12 months later. The primary aim of the study is to compare the effects of ISTS and UC on post-concussive symptoms and emotional distress at the 6-month assessment. The investigators predict that participants who receive ISTS will report lower levels of post-concussive symptoms and emotional distress at the 6-month assessment. Secondary aims include comparing the longer term effects of ISTS and UC at the 12-month assessment, as well as comparing their effects on other outcomes such as post-traumatic stress symptoms, quality of life, resilience, and work activity.

ELIGIBILITY:
Inclusion Criteria:

1. Active military or National Guard/Reserve status
2. Enrollment within 2 years of return from Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) theater and subsequent operations.
3. Positive response to screening at post-deployment examination and positive response to questions 1,2, or 6 on the "2 + 10 Traumatic Brain Injury (TBI) Screening Questionnaire" or positive response to questions 1c, 4,5, or 6 on the Military Acute Concussion Evaluation (which corresponds to the critical sections of the Centers for Disease Control operational definition of Mild Traumatic Brain Injury (MTBI))
4. Has access to a telephone.

Exclusion Criteria:

1. Moderate or severe TBI (Glasgow Coma Scale < 13) requiring hospitalization
2. Active psychotic disorder (including schizophrenia and schizoaffective disorder), severe depression with active suicidal ideation at TBI clinic visit, or current bipolar disorder by history.
3. Enrollment into intensive treatment at TBI programs at Madigan or Womack Army Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2011-06; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rivermead Post Concussion Symptoms Questionnaire | 6 months
  16-item self-report measure of symptoms that commonly occur following head injury
Brief Symptom Inventory - 18 Global Severity Index | 6 months
  18-item self-report measure of emotional distress; the Global Severity Index includes all items which capture anxious, depressive, and somatic symptoms

SECONDARY OUTCOMES:
Effects on functioning, quality of life, pain, sleep, depression, posttraumatic stress, resilience, work activity, and health services usage. | 6 months
  Comparison of effects using the EuroQol, Patient Health Questionnaire-9 (PHQ-9), PTSD Checklist- Pittsburgh Sleep Quality Index (PSQI), 10-item Connor-Davidson Resilience Scale (CD-RISC), the Brief Inventory for Functioning Evaluation (B-IFE), and Cornell Services Index (CSI).
Effect of ISTS in demographic subgroups | 12 months
  Attention to minority versus non-minority racial and ethnic populations, and active duty military versus National Guard/Reserve populations.
Satisfaction with ISTS by participants and significant others | 12 months
  Evaluation of satisfaction with ISTS using Client Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Bell, MD, Principal Investigator — University of Washington; Nancy Temkin, PhD, Study Director — University of Washington
Locations (4):
- United States (4):
  - Duke University, Durham, North Carolina
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Madigan Army Medical Center, Fort Lewis, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Bell KR, Fann JR, Brockway JA, Cole WR, Bush NE, Dikmen S, Hart T, Lang AJ, Grant G, Gahm G, Reger MA, St De Lore J, Machamer J, Ernstrom K, Raman R, Jain S, Stein MB, Temkin N. Telephone Problem Solving for Service Members with Mild Traumatic Brain Injury: A Randomized, Clinical Trial. J Neurotrauma. 2017 Jan 15;34(2):313-321. doi: 10.1089/neu.2016.4444. Epub 2016 Oct 13. PMID 27579992